CLINICAL TRIAL: NCT00131482
Title: A Double-blind, Randomized, Placebo-controlled Phase 2b Study to Establish the Effective Dose Range and to Evaluate the Safety of Chrysalin in Adult Subjects With a Fractured Distal Radius
Brief Title: A Study to Evaluate the Safety and Effectiveness of Different Doses of Chrysalin in Adults Who Have a Broken Wrist
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Treatment with Chrysalin did not demonstrate benefit compared to placebo.
Sponsor: Capstone Therapeutics (Industry)
Responsible Party: Denise Lamon, Director, Regulatory Affairs, Capstone Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OL-ADRFX-03
Record Dates: First submitted 2005-08-16; First posted 2005-08-18 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Radius Fracture
Keywords: Chrysalin; TP508; Fracture; Wrist; Healing
MeSH Terms: conditions — Radius Fractures; Fractures, Bone | interventions — rusalatide acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 10 micrograms (Experimental)
  Interventions: Drug: Chrysalin
- 30 micrograms (Experimental)
  Interventions: Drug: Chrysalin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 3 micrograms (Experimental)
  Interventions: Drug: Chrysalin
- 1 microgram (Experimental)
  Interventions: Drug: Chrysalin

INTERVENTIONS:
Drug: Chrysalin — Patients were treated with a single percutaneous injection of Chrysalin 3 micrograms at the fracture site at the time of surgery.
  Arms: 3 micrograms
Drug: Chrysalin — Patients were treated with a single percutaneous administration of Chrysalin 1 microgram at the fracture site at the time of surgery.
  Arms: 1 microgram
Drug: Chrysalin — Patients were treated with a single percutaneous administration of Chrysalin 10 micrograms at the fracture site at the time of surgery.
  Arms: 10 micrograms
Drug: Chrysalin — Patients were treated with a single percutaneous administration of Chrysalin 30 micrograms at the fracture site at the time of surgery.
  Arms: 30 micrograms
Drug: Placebo — Patients were treated with a single percutaneous administration of placebo at the fracture site at the time of surgery.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety of Chrysalin, also known as TP508, and to determine the effectiveness of four doses of Chrysalin for treating broken wrists in adults.

DETAILED DESCRIPTION:
There is a medical need for a product that is safe and can accelerate the rate of bone healing, leading to a reduction in immobilization time. Chrysalin, also known as TP508, is a synthetic peptide (protein) that is an exact copy of part of the human protein thrombin, which is a protein that occurs naturally in the body. Chrysalin can be used to mimic part of the thrombin response after injury without stimulating any of the events associated with blood clotting, and can therefore accelerate the normal process of healing.

ELIGIBILITY:
Inclusion Criteria:

* An unstable and/or displaced fracture of the distal radius
* Fracture classified as primary intra-articular or extra-articular
* Male, or non-pregnant, non-lactating female at least 18 years old. If female of childbearing potential, must have confirmed negative pregnancy test prior to administration of study product. Must agree to use a medically approved method of birth control for 6 months.
* Need ability to understand study requirements, provide written informed consent, and comply with study protocol
* Need ability to understand and provide written authorization for use and disclosure of health information per Health Insurance Portability and Accountability Act (HIPAA)

Exclusion Criteria:

* History of distal radius fracture of the affected limb 2 years prior to study enrollment
* History of uncontrolled Type I or Type II diabetes mellitus
* History or clinical evidence of any active medical disease or condition which would make the subject, in the opinion of the investigator, unsuitable for the study, or could potentially confound the results of the study
* Concurrent use of other investigational (non-Food and Drug Administration [FDA]-approved) agent or device
* Participation in any other clinical study within 90 days prior to treatment with the study drug
* Female subjects who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2004-11; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Time to removal of all rigid immobilization for fracture | Assessed Weeks 1-8, and Weeks 10, 12 and 26 after treatment

SECONDARY OUTCOMES:
Time to clinical healing of the fracture | Assessed Weeks 1-8, and Weeks 10, 12 and 26 after treatment
Time to radiographic healing of the fracture | Assessed Weeks 1-8, and Weeks 10, 12 and 26 after treatment
Assessment of range of motion relative to unbroken wrist | Assessed Weeks 1-8, and Weeks 10, 12 and 26 after treatment
Assessment of grip strength relative to unbroken wrist | Assessed Weeks 1-8, and Weeks 10, 12 and 26 after treatment
Results of patient questionnaires | Questionnaires given Weeks 4, 6, 8, 10,12 and 26 after treatment
Incidence of treatment-emergent adverse events | Weeks 1-8, and Weeks 10, 12, 26 and 52 after treatment
Chemistry and hematology laboratory evaluations | Within 24 hours, and at Weeks 2, 4, 8, and 26 after treatment

CONTACTS AND LOCATIONS:
Overall Officials: James Ryaby, Ph.D., Study Chair — Capstone Therapeutics
Locations (1):
- OrthoLogic, Tempe, Arizona, United States